CLINICAL TRIAL: NCT03155555
Title: Comparison of Carotid Peak Systolic Velocity Variation With Aortic Peak Systolic Velocity Variation in Pediatric Non-Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Subhrashis Guha Niyogi, Junior Resident, Department of Anaesthesia and Intensive care, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/3046/MD/400
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia, General; Anesthesia, Endotracheal; Mechanical Ventilation; Fluid Responsiveness
Keywords: Fluid Responsiveness; Pediatric surgery; General endotracheal anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Children aged 1-12 years undergoing major surgeries under general endotracheal anaesthesia with mechanical ventilation under neuromuscular blockade
  Interventions: Other: Measurement of aortic and carotid Doppler peak systolic velocity variation

INTERVENTIONS:
Other: Measurement of aortic and carotid Doppler peak systolic velocity variation — Aortic peak systolic velocity variation to be measured by echocardiography from apical five chamber and suprasternal windows alongwith carotid peak systolic velocity variation by Doppler ultrasound simultaneously at intermittent time points intermittently.

SUMMARY:
The purpose of this study is to evaluate whether carotid Doppler peak systolic velocity can be an easy to measure possible surrogate for echocardiographic measurement of aortic peak systolic velocity variation which is an index of fluid responsiveness in mechanically ventilated children intra-operatively.

ELIGIBILITY:
Inclusion Criteria:

• Patients scheduled for mon-cardiac surgeries under general endotracheal anaesthesia in supine position with expected duration more than 1 hour

Exclusion Criteria:

* Known congenital heart disease
* Any non-sinus rhythm, arrhythmias
* Patients on vasoactive medications
* Chest wall deformities, situs non solitus (eg. dextrocardia)
* Patients scheduled for open chest surgeries
* History of neck surgery/ carotid interventions

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible patients consenting for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Comparison of carotid peak systolic velocity variation with aortic peak systolic velocity variation | Measurements made within 3 minutes
  Comparison of carotid peak systolic velocity variation with aortic peak systolic velocity variation by Bland-Altman analysis

SECONDARY OUTCOMES:
Correlation between aortic peak systolic velocity variation measured from apical and suprasternal windows | Measurements made within 3 minutes
  Correlation between aortic peak systolic velocity variation measured from apical and suprasternal windows by Bland-Altman analysis

CONTACTS AND LOCATIONS:
Overall Officials: Subhrashis Guha Niyogi, MBBS, Principal Investigator — Junior Resident
Locations (1):
- Postgraduate Institute of Medical Education & Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niyogi SG, Sen IM, Jayant A, Mandal B, Bhardwaj N, Yaddanapudi S, Mathew P. Surrogate indices of aortic peak systolic velocity variation to monitor fluid responsiveness in pediatric non-cardiac surgery: a prospective observational study. J Clin Monit Comput. 2020 Dec;34(6):1159-1166. doi: 10.1007/s10877-019-00431-8. Epub 2019 Dec 7. PMID 31811550